CLINICAL TRIAL: NCT01283698
Title: An Investigator-blind, Controlled Study to Assess the Efficacy of Distinct Combinations of LAS 41004 in Different Concentrations Compared to Placebo and to Active Control in a Psoriasis-Plaque-Test
Brief Title: Clinical Trial to Investigate Efficacy of LAS41004 in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H553000-1005; 2010-022281-27 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Psoriasis
Keywords: psoriasis; topical; PPT
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- LAS 41004 dosage 1 (Experimental): dosage 1, once daily
  Interventions: Drug: Experimental: LAS 41004 dosage 1
- LAS 41004 dosage 2 (Experimental): dosage 2, once daily
  Interventions: Drug: Experimental: LAS 41004 dosage 2
- LAS 41004 dosage 3 (Experimental): dosage 3, once daily
  Interventions: Drug: Experimental: LAS 41004 dosage 3
- placebo (Placebo Comparator): once daily
  Interventions: Drug: Placebo Comparator: placebo
- Reference (Active Comparator): once daily
  Interventions: Drug: Reference

INTERVENTIONS:
Drug: Experimental: LAS 41004 dosage 1 — dosage 1, once daily
  Arms: LAS 41004 dosage 1
Drug: Experimental: LAS 41004 dosage 2 — LAS 41004 dosage 2, once daily
  Arms: LAS 41004 dosage 2
Drug: Experimental: LAS 41004 dosage 3 — dosage 3, once daily
  Arms: LAS 41004 dosage 3
Drug: Placebo Comparator: placebo — once daily
  Arms: placebo
Drug: Reference — Active Comparator,once daily
  Arms: Reference

SUMMARY:
The aim of the study is to intra-individually compare the dose-related efficacy of LAS41004 in a Psoriasis Plaque Test (PPT)

ELIGIBILITY:
Inclusion Criteria:

* • Male or female patients between 18 and 75 years of age with a diagnosis of stable plaque-type psoriasis (psoriasis vulgaris) for at least 6 month

  * Psoriasis plaques that are suitable to be defined as target area lesions by the following criteria:

    * Psoriasis plaques must be located at trunk and/or extremities. Plaques that are located on the head (incl. scalp), palms, sole of the feet, intertriginous or genitoanal areas are not suitable as target areas
    * Comparable psoriasis plaques with at least "2" in each score (Range 0-4) for the three distinct symptoms scaling; erythema; and induration
    * No more than 3 points difference in total score (= sum of scores for scaling, erythema and induration; Range 0-12) of the chosen comparable psoriasis plaques
    * Enough psoriatic surface area to define 5 clearly distinguishable (minimum distance between test areas: 1cm) test areas of at least 1 cm² plaque size
  * Patient is willing and able to comply with the requirements of the clinical study protocol. In particular, patient must adhere SCIderm GmbH Confidential Almirall Hermal GmbH Study protocol EudraCT No. 2010-022281-27 Protocol No. H553000-1005 Version 1.0 to concomitant therapy prohibitions of the test areas and must agree to avoid intense UV exposure of the test areas during the study
  * Written informed consent to participate in the study, prior to any study related procedures, indicating an understanding of the purpose of the study
  * A patient of childbearing potential agrees to use one of the following contraceptive methods for the duration of the study and the following 4 weeks after the end of study :

    * Strict abstinence (exception: male partner with a vasectomy for at least 3 months prior to study entry is allowed)
    * Combined oral, implanted or injectable contraceptives on a stable dose for at least 3 months prior to study entrance
    * Intrauterine device (IUD) inserted for at least 1 month prior to study entrance

Exclusion Criteria:

* Too few body surface area covered with psoriasis plaques that meet the specified inclusion criteria to be defined as 5 clearly distinguishable test areas
* Any condition that may interfere with the study assessments or sonographic measurements of the skin and/or may have an influence on skin immune response (incl. open wounds)
* Known adverse reactions of any severity or hypersensitivity to any ingredient of the test products
* No willingness to avoid induction of heavy sweating, e.g. due to sauna visits, excessive sports activities during the study course
* No willingness to avoid swimming, bathing or wetting of the designated test areas between visits
* Pregnant or breast-feeding women
* A medical condition that may put the patient at a general risk and therefore would prevent participation in the clinical trial (including but not limited to: serious infectious diseases, major surgery within the last 4 weeks, coronary artery disease, renal impairment, hepatic impairment, uncontrolled metabolic diseases, disorders of the calcium metabolism, autoimmune diseases)
* History or presence of malignant disease (other than surgically removed basal cell carcinoma) and/or auto immune diseases
* Current diagnosis of guttate, erythrodermic or pustular psoriasis
* Patients who did not respect the following wash-out periods prior or during the study:

Treatment Wash out period Topical treatment in the test area Any topical anti-psoriatic drug 2 weeks Systemic treatment Biologics 6 months Any other systemic treatment (corticosteroids, ciclosporin, MTX, fumaric acid esters) 3 months Procedures Phototherapy 4 weeks

* Significant skin diseases other than plaque-type psoriasis (psoriasis vulgaris), incl. skin infections
* Excessive sunlight exposure within 28 days prior to study entry and during the conduct of the study
* Usage of any topical formulation (incl. cosmetics, emollients, etc) on the designated target areas during the course of the study
* Vaccination 6 days prior to enrolment or during the study
* Subjects who are - in the opinion of the investigator - unreliable, and/or non-compliant, and/or who present with any condition or treatment (including cosmetic products) that may interfere with psoriasis or the conduct of the trial
* Participation in any other clinical trial within 30 days prior or during this trial
* Subject is an adult under guardianship, hospitalised, deprived of freedom or unable to communicate or cooperate with the investigator due to language or mental problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Decrease in thickness of infiltration | 15 days
  measurement will be performed by ultrasound, comparing data from baseline (day1) vs end of trial (day15)

SECONDARY OUTCOMES:
Change in clinical score | 15 days
  scoring will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Change in erythema score | 15 days
  scoring will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Change in Induration score | 15 days
  scoring will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Change in Scaling score | 15 days
  scoring will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Number of skin reactions per patient as a measure of safety and tolerability | 15 days
  daily scoring will be performed by investigator
Number of AEs per patients as a measure of safety and tolerability | 15 days
  reporting will be performed by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (1):
- Almirall Investigational Sites#1, Mahlow, Germany